CLINICAL TRIAL: NCT03383406
Title: A Phase II Trial of Ifosfamide, Etoposide, Cytarabine, and Methotrexate (IVAM) Chemotherapy for Refractory or Relapsed Diffuse Large B Cell Lymphoma
Acronym: IVAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AsanMC_LMP2017-001
Record Dates: First submitted 2017-10-30; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Ifosfamide; Etoposide; Cytarabine; Methotrexate; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I Ifosfamide, Etoposide, Cytarabine, and Methotrexate (IVAM) (Experimental)
  Interventions: Drug: Ifosfamide, Etoposide, Cytarabine, and Methotrexate (IVAM) Chemotherapy

INTERVENTIONS:
Drug: Ifosfamide, Etoposide, Cytarabine, and Methotrexate (IVAM) Chemotherapy — Every cycle(4weeks)
  Subject will receive Ifosfamide 1.5 g/m2 over 2 hours for Day1~Day5 by Intravenous infusion, Etoposide 150 mg/m2 over 3 hours on Day1~Day3 by Intravenous infusion, Cytarabine 100 mg/m2 over 1 hour on Day1~Day3 by Intravenous infusion.
  Other Names: IVAM

SUMMARY:
A phase II trial of ifosfamide, etoposide, cytarabine, and methotrexate (IVAM) chemotherapy for refractory or relapsed diffuse large B cell lymphoma

DETAILED DESCRIPTION:
Diffuse Large B-Cell lymphoma is currently used as a standard treatment, with a combination of chemotherapy (R-CHOP), which includes Rituximab. However, the survival rate is very poor if the primary treatment is refractory or relapsed within a year or less. The duration of these patients ' lives is around one year and the five-year survival rate is 15-20 %. Thus, a new treatment strategy is needed to improve the survival of the patient with DLBCL, which are either refractory and relapsed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed adult patients diagnosed with DLBCL refractory or relapsed.
* Large scale B cell lymphoma not received ASCT(autologous stem-cell transplantation ) after primary chemotherapy
* At least one measurable lesion

  * ≥1 cm in greatest transverse diameter by spiral CT
  * ≥2 cm in greatest transverse diameter by conventional CT
  * ≥1 cm in visible skin lesion
  * ≥2 cm in digital exploration
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2.
* Age 19~59yrs
* MUGA(multiple gated acquisition scan ): Non-Clinical significant and 2D-Echo( Cardiac Index ≥ 50 % )
* Adequate renal function: serum creatinine level < 2.0 mg/dL(177μmol/L) Adequate liver functions: Transaminase (AST/ALT) < 3 X upper limit of normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver), bilirubin < 2 X upper normal value (or < 5 x upper limit of normal in the presence of DLBCL involvement of the liver)
* Adequate hematological function: hemoglobin ≥ 9.0 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL,
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.

Exclusion Criteria:

* Pre-treatment for ASCT
* Central nervous system (CNS) involvement by lymphoma
* Prior history of malignancies other than lymphoma (except for treated Non Melanoma Skin Cancer, early gastric cancer or carcinoma in situ of the cervix or breast or untreated prostatic cancer without any plan for a treatment) unless the patient has been free of the disease for ≥ 5 years
* Pregnant or lactating woman, Childbearing potential not employing adequate contraception
* Active uncontrolled infections(Bacterial, Viral, Fungus)
* Other serious illness or medical conditions
* Other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response | 2 to 3 weeks after completion of the 2nd cycle of treatment (each cycle is 28 days)
  CT, PET-CT(positron emission computed tomography )

SECONDARY OUTCOMES:
Assess response rate | 4 to 5 weeks after completion of the 4th cycle of treatment(each cycle is 28 days)
  CT, PET-CT
Assess response rate | 6 to 8 weeks after completion of the 6th cycle of treatment(each cycle is 28 days)
  CT, PET-CT
Assess response rate | After completion of the treatment, up to 24weeks
  CT, PET-CT
Assess response rate | After 1year completion of the treatment up to 1year
  CT, PET-CT
Assess response rate | Afer 2years completion of the treatment up to 3years
  CT, PET-CT

OTHER OUTCOMES:
Assess overall survival | The time from the 1st day of treatment to death of any cause or the date of last follow-up, assessed up to 66 months
  CT, PET-CT

IPD SHARING:
Plan to Share IPD: Undecided